CLINICAL TRIAL: NCT06555419
Title: An Open Label, Single Cohort Study to Assess the Pharmacokinetic Profile of Nusinersen (BIIB058) Administered Via the ThecaFlex DRx™ System (PIERRE-PK)
Brief Title: A Study to Find Out How Nusinersen is Processed in the Body When Given Through the ThecaFlex DRx™ System in Adult and Pediatric Participants With Spinal Muscular Atrophy (PIERRE-PK)
Acronym: PIERRE-PK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Alcyone Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 295SM101; 2024-514239-21-00 (Other: EU CTIS Number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nusinersen Via LP and ThecaFlex DRx System (Experimental): Participants will receive a maintenance dose of nusinersen, 12 milligrams (mg) via LP in the PIERRE-PK study, followed by implantation of the ThecaFlex DRx System and the subsequent nusinersen 12 mg maintenance dose via the system in the PIERRE study.
  Interventions: Drug: Nusinersen; Device: ThecaFlex DRx System

INTERVENTIONS:
Drug: Nusinersen — Administered as specified in the treatment arm.
  Other Names: BIIB058
Device: ThecaFlex DRx System — Implanted as specified in the treatment arm.

SUMMARY:
In this PIERRE-PK study, researchers will learn how the body processes nusinersen when it is given through the ThecaFlex DRx™ System, compared to when nusinersen is given by lumbar puncture (LP). The ThecaFlex DRx system is an investigational implantable medical device developed by Alcyone Therapeutics, Inc. It consists of a catheter, which is a flexible tube, connected to a port which is placed under the skin. Alcyone Therapeutics, Inc. has an ongoing study called PIERRE to test the ThecaFlex DRx system. Participants with spinal muscular atrophy (SMA) in the PIERRE study may be enrolled in the PIERRE-PK study.

The main objective of the PIERRE-PK study is to learn how the body processes nusinersen when given by the ThecaFlex DRx system compared to a lumbar puncture. The main questions researchers want to answer are:

* What is the highest amount of nusinersen found in the blood after dosing?
* How much nusinersen is found in the blood over the first 24 hours after dosing?

The PIERRE-PK study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 30 days for this study and may overlap with the PIERRE study.
* Participants will receive a dose of nusinersen by lumbar puncture.
* The ThecaFlex DRx system will be implanted after the lumbar puncture, as part of the PIERRE study.
* Participants will receive a dose of nusinersen by the ThecaFlex DRx system, as part of the PIERRE study.
* Researchers will take blood samples before and after each dose. The last blood sample will be taken 24 hours after the dose.
* The total study duration for each participant in the PIERRE-PK study will be approximately 5 months. This period will overlap with the participant's first 5 months in the PIERRE study.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the Pharmacokinetic (PK) profile of nusinersen delivered via standard LP and via the ThecaFlex DRx System in participants with SMA.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is on regular maintenance dosing of nusinersen (12 milligrams [mg] dose) every 4 months, with 4 months (± 2 weeks) between the LP-delivered study dose and the last nusinersen dose prior to study enrollment.
* Participants must be enrolled in the PIERRE study to be eligible for enrolment in the PIERRE PK study.

Key Exclusion Criteria:

* Ongoing participation or participation within 6 months or 5 half-lives of the agent (whichever is longer) of enrollment in other interventional clinical trials for the treatment of SMA (except for the PIERRE study or interventional clinical trials of myostatin inhibitors [e.g., apitegromab and taldefgrobep alfa]).
* Participant is naïve to nusinersen treatment.
* Participant is receiving nusinersen at a dose other than 12 mg.
* Participant has already undergone implantation of the ThecaFlex DRx system.
* Participant is pregnant, currently breastfeeding, or intending to become pregnant during the study.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Nusinersen Delivered via Standard LP and via ThecaFlex DRx System | Pre-dose and at multiple time points post-dose up to 4 months
Area Under the Plasma Concentration-Time Curve From Zero Time to 24 Hours After Intrathecal Administration (AUC0-24h) of Nusinersen Delivered via Standard LP and via ThecaFlex DRx System | Pre-dose and at multiple time points post-dose up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- United States (10):
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center | Department of Neurology_Palo Alto, Palo Alto, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospita, Grand Rapids, Michigan
  - Milton S. Hershey Medical Center | Pennsylvania State University_Hershey, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Childrens Hospital Houston, Houston, Texas
  - Stacey Hall Developmental Pediatrics, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters_Norfolk, Norfolk, Virginia
- Hôpital Raymond Poincaré, Garches, Hauts De Seine, France
- Universitaetsklinikum Essen, Essen, Germany
- Italy (2):
  - Fondazione Serena Onlus - Centro Clinico Nemo_Milano, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Poland (2):
  - Szpital Specjalistyczny im. L.Rydygiera w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe_Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/